CLINICAL TRIAL: NCT01725568
Title: Master Study of the Implantable Cardiac Monitor "BioMonitor"
Brief Title: BioMonitor Master Study
Acronym: BioMonitor
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: 60
Record Dates: First submitted 2012-11-06; First posted 2012-11-14 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: ATRIAL FIBRILLATION, Syncope
MeSH Terms: conditions — Atrial Fibrillation; Syncope

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Implantable cardiac monitor diagnostics: Patients has standard indication for implantable cardiac monitor diagnostic.
  Interventions: Device: BioMonitor

INTERVENTIONS:
Device: BioMonitor — Implantable cardiac monitor

SUMMARY:
The BioMonitor is an implantable cardiac monitor used to automatically detect and record episodes of arrhythmia in patients with bradycardia, tachycardia, asystole and atrial fibrillation. The study will be conducted to support regulatory approvals outside of Europe. This BioMonitor Master study is designed to investigate the clinical efficacy and safety of the BioMonitor.

ELIGIBILITY:
Inclusion Criteria:

* Suspected cardiac arrhythmia OR Previous AF diagnosis OR AF diagnosis before or after ablation procedure OR Stroke of unknown origin.

Exclusion Criteria:

* Implanted ICD or cardiac pacemaker
* Allergy to patch electrodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with standard ICM indication who are referred to the hospital
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2012-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
SADE free-rate | at 3 month follow-up
  SADE free-rate > 90% at 3 month follow-up
Rate of appropriate QRS detection | at 6 week follow-up
  Rate of appropriate QRS detection > 90% (based on comparison with Holter ECG recording)

OTHER OUTCOMES:
Sensitivity and Positive Predictive of episode detection | 1 year
  Sensitivity and Positive Predictive Value of each automatically detected cardiac arrhythmia that was stored as subcutaneous electrocardiogram by the BioMonitor (6 week, 3 and 12 month follow-up data)
Adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dietmar Baensch, Professor, Principal Investigator — University of Rostock, Germany
Locations (1):
- University of Rostock, Rostock, Germany